CLINICAL TRIAL: NCT02943499
Title: Mechanisms of Mindfulness for Smoking Cessation: Optimizing Quantity and Quality.
Brief Title: Mechanisms of Mindfulness for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Judson Brewer, Principal Investigator, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1R61AT009337-01 (NIH)
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Comparator App/Training (Active Comparator): This is a standard smoking cessation smartphone app using the latest evidence-based smoking cessation methods and behavior change theory. Subjects will be encouraged to set a quit date of 3 weeks, to allow comparison to experimental arm quit date.
  Interventions: Behavioral: App/Training; Device: Smartphone
- Experimental App/Training (Experimental): This is a 3-week smartphone-based training program that trains mindfulness for smoking cessation by helping smokers self-monitor their smoking habits, recognize when and how often they smoke, identify triggers for smoking, and learn methods to become more mindful of triggers, to quit smoking with a target quit date of 3 weeks.
  Interventions: Behavioral: App/Training; Device: Smartphone

INTERVENTIONS:
Behavioral: App/Training — This is a free smoking cessation smartphone app using the latest evidence-based smoking cessation methods and behavior change theory. The app allows users to set a quit date, financial goals, and reminders, track daily smoking habits with an easy-to-use calendar, see graphs tracking money saved and number of packs not smoked, receive health milestones and craving tips to stay motivated, connect with social networks to give milestone updates, create a video diary, and watch personalized video messages from loved ones
  Arms: Active Comparator App/Training
Behavioral: App/Training — It is comprised of twenty-two modules of 10-15 minutes each, designed to teach mindfulness for smoking cessation using psychoeducation-based audio and videos, animations to reinforce key concepts, and in vivo exercises. In addition, 5 bonus modules become available upon completion of earlier modules; these may be accessed for additional practices to bolster other modules.
  Arms: Experimental App/Training
Device: Smartphone

SUMMARY:
The purpose of this study is to understand brain mechanisms of app-based mindfulness training in smokers ages 21 to 65 years.

ELIGIBILITY:
Inclusion Criteria:

* 21-65 years of age
* Smoke 10+ cigarettes/day
* < 3 months abstinence in the past year
* Have a smartphone; and motivated to quit smoking
* Score >18 of 20 on Action subscale of the Readiness to Change Questionnaire

Exclusion Criteria:

* Any usage of psychotropic medication: not on a stable dosage 6+ months
* Prior participation in a mindfulness course or regular meditation practice (>20 min/week)
* Serious psychiatric, cognitive, or medical disorder
* MRI contraindications
* Structural brain damage as well as other brain abnormalities revealed by the MRI
* Claustrophobia
* Not being fluent in English
* Recreational drug use
* Pregnant women
* History of a neurological disorder
* Current participation in a smoking study
* Adults unable to consent
* Prisoners

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-10; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts, Worcester, Worcester, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator App/Training: This is a standard smoking cessation smartphone app using the latest evidence-based smoking cessation methods and behavior change theory. Subjects will be encouraged to set a quit date of 3 weeks, to allow comparison to experimental arm quit date.
  App/Training: This is a free smoking cessation smartphone app using the latest evidence-based smoking cessation methods and behavior change theory. The app allows users to set a quit date, financial goals, and reminders, track daily smoking habits with an easy-to-use calendar, see graphs tracking money saved and number of packs not smoked, receive health milestones and craving tips to stay motivated, connect with social networks to give milestone updates, create a video diary, and watch personalized video messages from loved ones
  Smartphone
- Experimental App/Training: This is a 3-week smartphone-based training program that trains mindfulness for smoking cessation by helping smokers self-monitor their smoking habits, recognize when and how often they smoke, identify triggers for smoking, and learn methods to become more mindful of triggers, to quit smoking with a target quit date of 3 weeks.
  App/Training: It is comprised of twenty-two modules of 10-15 minutes each, designed to teach mindfulness for smoking cessation using psychoeducation-based audio and videos, animations to reinforce key concepts, and in vivo exercises. In addition, 5 bonus modules become available upon completion of earlier modules; these may be accessed for additional practices to bolster other modules.
  Smartphone
Period: Overall Study
Arm/Group | Active Comparator App/Training | Experimental App/Training
Started | 41 | 39
Completed | 34 | 34
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Population: 1 individual was excluded from analysis in the experimental app/training arm because they did not meet MRI inclusion criteria at follow-up
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator App/Training | Experimental App/Training | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 33 | 67
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (11) | 46 (11) | 45 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 45
  Male | 9 | 13 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 32 | 31 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 33 | 31 | 64
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
PCC reactivity [Mean (Standard Deviation); unit: BOLD signal] — Smoking cue reactivity in the posterior cingulate cortex (PCC) as measured by blood oxygen-level dependent (BOLD) response
  BOLD signal | 18.9 (22.2) | 22.2 (21.6) | 20.5 (22)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Blood Oxygen Level Dependent (BOLD) Signal
Description: BOLD signal change will be measured by fMRI and analyzed using statistical parametric mapping
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: BOLD signal
Arm/Group | Active Comparator App/Training | Experimental App/Training
Number analyzed (Participants) | 34 | 33
BOLD signal | 16.1 (23.4) | 18.6 (22.2)
Statistical Analysis 1: Comparison: Active Comparator App/Training vs Experimental App/Training; To examine between-group differences in pre- vs. post-treatment cue reactivity, the post-treatment PCC BOLD response for the smoking vs neutral contrast was subtracted from the baseline response. The groups were then compared directly on this measure using a t-test; Test type: Superiority; p = 0.92, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Active Comparator App/Training | Experimental App/Training
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/33
Other Adverse Events (participants affected / at risk) | 1/34 | 2/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Comparator App/Training (N=34) | Experimental App/Training (N=33)
Prolapse of the mitral and tricuspid valves (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Comparator App/Training (N=34) | Experimental App/Training (N=33)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ear infection (Ear and labyrinth disorders) | 0 | 1
Back injury (Musculoskeletal and connective tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
There are several limitations, including the short duration of follow up for smoking outcomes and the specific focus on a single region of interest.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT02943499/Prot_SAP_000.pdf